CLINICAL TRIAL: NCT05381298
Title: Biological Evaluation of Indirect Restorations in Endodontically-treated Posterior Teeth With Deeply Located Proximal Margins Following Deep Margin Elevation Versus Surgical Crown Lengthening: A Randomized Controlled Trial
Brief Title: Deep Margin Elevation Vs Crown Lengthening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Tarek Farouk, principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19750
Record Dates: First submitted 2022-05-12; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Margin Elevation (Experimental)
  Interventions: Procedure: Deep Margin Elevation using resin composite; Procedure: Surgical Crown Lengthening
- Surgical Crown Lengthtening (Experimental)
  Interventions: Procedure: Deep Margin Elevation using resin composite; Procedure: Surgical Crown Lengthening

INTERVENTIONS:
Procedure: Deep Margin Elevation using resin composite — After completion of the root canal treatment of the offended tooth and comprehensive evaluation of the obtained treatment, the randomly allocated patients will undergo deep margin elevation procedure where rubber dam isolation will be accomplished Followed by proper matricing and wedging ) followed by selective enamel etching for 10 seconds then universal adhesive application following the manufacturer instructions followed by application of flowable resin composite for the first 1 mm and light cured for 20 seconds according to the manufacturer recommendations followed by application of packable bulk fill composite to elevate the margins and light cured following the manufacturer instructions.
Procedure: Surgical Crown Lengthening — Participants in this group will undergo surgical crown lengthening in which an internal bevel incision will be done buccally and lingually followed by full thickness flap reflection using mucoperiosteal elevator, then interproximal bone removal will be done using end cutting bur to the planned position away from the margins by 3 mm. The flap will be displaced apically with apically positioned sutures. Postoperative instructions will be given to the patient aiming to control postsurgical complications including pain and swelling. Suture removal and assessment of the surgical site will be done after two weeks

SUMMARY:
The present clinical trial will be conducted to reject or accept the null hypothesis that in endodontically treated posterior teeth with deeply located proximal margins, will the Deep Margin Elevation will have better results from surgical crown lengthening in terms of biological criteria?

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent endodontic treatment in the posterior region
* 18-40 years
* Male and Females
* Medically free patients
* Patients with healthy periodontium
* Patients with thick biotype.
* Patients having proximal margins violating the biological width

Exclusion Criteria:

* Patients with chronic periodontal disease.
* Patients with persistent poor oral hygiene.
* Patients with unsuccessful root canal treatment.
* Periapical Abscess or Fistula.
* Patients with proximal margins beyond the bone level.
* Patients with developmental dental anomalies.
* Patients undergoing or will start orthodontic treatment
* Patients with removable prosthesis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 12 month
  the clinical attachment level will be measured from restoration margin to the base of the clinical gingival sulcus according to Günay et al

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided